CLINICAL TRIAL: NCT05428852
Title: Keto-Brain: Investigating the Use of Ketogenic Diets in Brain Metastases
Brief Title: Keto-Brain:Investigating the Use of Ketogenic Diets in Brain Metastases
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: IRB Approval Expiration
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Jeff Volek, Professor, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2020C0046; NCI-2023-10603 (Other: National Cancer Institute); OSU-19277 (Other: Ohio State University Comprehensive Cancer Center)
Record Dates: First submitted 2022-06-14; First posted 2022-06-23 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Brain Metastases, Adult
MeSH Terms: conditions — Brain Neoplasms | interventions — Mental Status and Dementia Tests; Diet Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of Care (Active Comparator): Patients receive standard of care therapy with SRS and AICR Diet education.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Neurocognitive Assessment; Other: Questionnaire Administration; Device: Fitbit
- Standard of Care + Ketogenic Diet (Experimental): (standard of care, ketogenic diet) Patients receive standard of care with SRS. Patients undergo a controlled feeding period ketogenic diet comprising of meals for the first week and then transition into a free living with guided support type of intervention.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Neurocognitive Assessment; Other: Questionnaire Administration; Device: Fitbit; Dietary Supplement: Dietary Intervention

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative Studies
Other: Neurocognitive Assessment — NRG-CC
Other: Questionnaire Administration — Ancillary studies
Device: Fitbit — Fitbit Activity Tracking
Dietary Supplement: Dietary Intervention — Undergo ketogenic diet
  Arms: Standard of Care + Ketogenic Diet

SUMMARY:
This pilot study will be a single center, randomized controlled study of 24 participants with diagnosed BM (various primary disease sites) comparing the effect of a ketogenic (n=12) and AICR (n=12) diet. Potential participants will be identified via medical record reviews and chart reviews. Eligibility of patients will be assessed via medical record review. Randomization will be balanced by blocks of random sizes but no stratification due to the small sample size. Both groups will undergo a 16-week diet intervention where research dietitians will provide educations, recipes and grocery lists on the participants assigned diet. Each group will receive 4-7 days worth of food prior to testing days to both aid in transitioning to each dietary arm and to ensure that the metabolic needs for each arm are met. In an effort to maintain a patient centric focus and monitor changes in quality of life (QOL) all patients will complete psychosocial and behavioral inventories. These inventories aim to capture a holistic view on the proposed nutritional intervention during treatment. Primary outcomes will be determined at baseline, 8 weeks, and 16 weeks while patient-centric outcomes will be assessed every four weeks. Participants will have counseling by the attending physician for additional applicable medications for any treatment related side effects or toxicities. The intervention groups will undergo their randomized dietary regimen for 16 weeks.

DETAILED DESCRIPTION:
Neurological tissues are among the most common (>10% of cancer patients) and debilitating sites for metastatic disease to develop. The brain is a 'sanctuary site' for many cancer cells and remains a challenging site to treat. Surgery and radiation therapies are the most common treatments. The investigators hypothesize that the metabolic adaptations associated with a well-formulated ketogenic diet that induces nutritional ketosis will significantly improve the response to surgery and radiation in patients with brain metastases. To date, numerous preclinical studies have demonstrated the ability of nutritional ketosis and caloric restriction to augment the therapeutic efficacy of radiotherapy. Use of a ketogenic diet is known to decrease the protein expression of HIF-1 and VEGFR2, and may increase radio sensitivity by normalizing tumor vasculature and increasing facilitated oxygen delivery to tumor cells. Several additional proposed mechanisms exist for enhancing radiosensitivity of the malignancy including: HDAC dependent mechanisms, ATP deprivation, mitochondrial ROS production and downregulation of IGF-1 receptor. Short-term fasting, a way to increase ketones acutely, has been demonstrated to speed up mitotic rates and thus facilitate a DNA damage sensitization. Lastly, a recent study showed that glucose restriction lowered Ki-67 expression, clonogenic frequency and rate of proliferation in gliomaspheres in vitro.

The investigating team team has an established expertise in conducting ketogenic diet interventions. Many individuals have adopted a low-carbohydrate diet for health reasons, yet there is scarce professional support available to provide guidance and support, especially for ketogenic diets. The investigators have scientific expertise and practical knowledge of both ketogenic and current standard of care cancer diets combined with a passion to empower people with the tools to implement these eating approaches into the participant's lifestyle. This project is highly patient-centered. The investigators will support patients who are randomized into either one of the intervention groups and provide them with a personalized eating plan designed to have maximal therapeutic impact and positively impact their lives. To that end, this project is unique in that it is highly patient-centered while also designed to have a substantial scientific and practical impact on medical management of brain metastasis treatments.

ELIGIBILITY:
Inclusion Criteria:

* Measurable brain lesions noted on baseline MRI imaging
* Graded Prognostic Assessment > 1.5
* Body mass index (BMI) ≥18 kg/m2
* Eastern Cooperative Oncology Group (ECOG) Performance status of 0-1 (0=participant has either normal activity, 1= participant has some symptoms but is nearly full ambulatory)
* Able and willing to follow prescribed diet intervention
* Scheduled to receive SRS

Exclusion Criteria:• Undergoing whole brain radiation therapy

* BMI <18 kg/m2
* Pregnant or nursing women
* Not willing to be randomized into either of the dietary interventions
* Unable to provide Informed Consent
* No previous diagnosis of small cell lung carcinoma
* No previous or suspected leptomeningeal disease
* Type 1 diabetes or insulin-dependent Type II diabetes
* Abnormal renal function (GFR < 55 mL/min, creatinine >2.0, urinary albumin >1 g/day) Not MRI eligible

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-09-26 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of maintaining a ketogenic versus AICR diet in patients with brain metastasis selected for radiosurgery | Up to 16 weeks
  Summaries from questionnaires will be plotted over time to assess adherence and compliance to the ketogenic diet.
Feasibility of maintaining a ketogenic diet in patients with brain metastasis selected for radiosurgery | Up to 16 weeks
  Summaries from ketone logs will be plotted over time to assess adherence and compliance to the ketogenic diet.
Metabolic outcomes of a ketogenic versus AICR diet in patients with brain metastasis selected for radiosurgery | Up to 16 weeks
  Summaries from blood markers will be plotted over time to assess adherence and compliance to the ketogenic diet.
Number of Participants with partial-or-complete response according to RECIST v1.1 | Baseline up to 16 weeks
  use a Chi-squared test for the association between treatment group and partial-or-complete response according to RECIST v1.1

SECONDARY OUTCOMES:
Preliminary effects of the ketogenic versus AICR diet on Neurocognitive Function Scores in BM individuals undergoing radiation therapy | Baseline up to 16 weeks
  same linear mixed effects model as for the primary objective, but with the following quality-of-life endpoints as outcomes
Preliminary effects of the ketogenic versus AICR diet on PROMIS Cognitive Function Short Form 8a Scores in BM individuals undergoing radiation therapy | Baseline up to 16 weeks
  same linear mixed effects model as for the primary objective, but with the following quality-of-life endpoints as outcomes
Preliminary effects of the ketogenic versus AICR diet on Heart Hope Scale in BM individuals undergoing radiation therapy to asses quality of life | Baseline up to 16 weeks
  same linear mixed effects model as for the primary objective, but with the following quality-of-life endpoints as outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Volek, PhD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu

DOCUMENTS (2):
  • Study Protocol (2022-04-13): https://cdn.clinicaltrials.gov/large-docs/52/NCT05428852/Prot_000.pdf
  • Informed Consent Form (2022-04-13): https://cdn.clinicaltrials.gov/large-docs/52/NCT05428852/ICF_001.pdf